CLINICAL TRIAL: NCT06635798
Title: A Multicentre, Randomized, Double-blind, Human Tetanus Immunoglobulin(HTIG) Controlled Phase III Clinical Trail to Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity Characteristics of GR2001 Injection for Indication of Prophylaxis Against Tetanus
Brief Title: A Phase III Clinical Trail to Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity Characteristics of GR2001 Injection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GR2001-002
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Tetanus
Keywords: Tetanus; Human Tetanus Immunoglobulin; GR2001 Injection
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GR2001 (Experimental): If randomized to GR2001, participant will receive a single IM gluteal injection of GR2001
  Interventions: Biological: GR2001
- HTIG (Active Comparator): If randomized to HTIG, participant will receive a single IM gluteal injection of HTIG
  Interventions: Biological: HTIG

INTERVENTIONS:
Biological: GR2001 — The packaging for GR2001 injection uses a borosilicate glass vial, a brominated halobutyl rubber stopper for injectable solutions and an aluminum-plastic combination cap for antibiotic vials as its primary packaging materials. The specification is 5mg/1ml per vial.
  Arms: GR2001
Biological: HTIG — The HTIG is a Chinese licensed Human Tetanus Immunoglobulin produced by Tonglu-Bio, which are derived from human plasma, and then purified and filled in the injectable vial form.
  Arms: HTIG

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of GR2001 injection with Human Tetanus Immunoglobulin(HTIG) in tetanus prophylaxis. Patients will receive either GR2001 injection or HTIG on study D0.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female adults aged ≥ 18 years；
2. Participants with suspected tetanus exposure (due to dirty or contaminated wounds from various injuries);
3. Participants who provide signed written informed consent form.

Exclusion Criteria:

1. Participants known to be allergic to the investigational medicinal product or those suffering from severe allergic conditions；
2. Suspect or diagnosed as tetanus;
3. Previously diagnosed as Immunoglobulin A (IgA) deficiency with anti-IgA antibodies；
4. Prior vaccination history of ≥ 3 doses of tetanus toxoid or tetanus toxoid- containing vaccine;
5. Females who are pregnant or with pregnancy test positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
The increase of anti-tetanus neutralizing antibody titers (∆ titers) | Baseline up to 12 hours after receipt of Investigational medicinal product.
  The proportion of participants with an increase of anti-tetanus neutralizing antibody titers (∆ titers) over protective level.

SECONDARY OUTCOMES:
The incidence of tetanus | Up to 105 days after receipt of Investigational medicinal product.
To evaluate the safety of GR2001 | Up to 105 days after receipt of Investigational medicinal product.
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0
To evaluate the peak plasma concentration(Cmax) of GR2001 | Up to 105 days after receipt of Investigational medicinal product.
To evaluate the Area under the plasma concentration versus time curve (AUC0-last,AUC0-inf) of GR2001 | Up to 105 days after receipt of Investigational medicinal product.
To evaluate the immunogenicity of GR2001 | Up to 105 days after receipt of Investigational medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanlin Wang, MD, Principal Investigator — Peking University People's Hospital; Zhanfei Li, MD, Principal Investigator — Tongji Hospital
Locations (20):
- China (20):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital Affiliated to Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Liuzhou Workers's Hospital, Liuchow, Guangxi
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Nanhua Hospital Affiliated to University of south China, Hengyang, Hunan
  - The Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang